CLINICAL TRIAL: NCT04067700
Title: Accuracy of Cardiopulmonary Exercise Testing in the Diagnosis of Myocardial Ischemia
Brief Title: CPET in Myocardial Ischemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Tomi Laitinen, Professor, chief physician, Kuopio University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5031365
Record Dates: First submitted 2019-08-22; First posted 2019-08-26 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Intervention Model Description: Patients who receive invasive coronary treatment will undergo additional coronary perfusion PET/CT and CPET tests six months after the treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Coronary perfusion PET/CT patients (Other)
  Interventions: Procedure: Invasive coronary treatment

INTERVENTIONS:
Procedure: Invasive coronary treatment — Coronary artery bypass surgery or percutaneous coronary intervention.

SUMMARY:
The investigators goal is to determine whether cardiopulmonary exercise testing (CPET) can be utilized in the diagnosis of myocardial ischemia. For the study participants the investigators will recruit patients who have been referred to myocardial perfusion PET/CT scan in Kuopio University Hospital. The participants will perform the CPET on a cycle ergometer on separate day after the perfusion scan. The investigators will compare the results of the PET/CT scan and CPET and evaluate if the possible perfusion defects detected in PET/CT correlate with the gas exchange parameters in CPET.

The patients who receive invasive coronary treatment (coronary bypass surgery or percutaneous coronary intervention) will be invited to perform additional CPET ja PET/CT tests six months after the treatment. The goal will be to determine whether the recovery of myocardial perfusion can be assessed with gas exchange parameters in CPET.

ELIGIBILITY:
Inclusion Criteria:

* Referral to coronary perfusion PET/CT scan in Kuopio University Hospital

Exclusion Criteria:

* Age under 18 years
* Pregnancy or breastfeeding
* Handicap
* Imprisonment
* Care under forensic psychiatry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-03 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Presence of myocardial ischemia assessed by the myocardial perfusion positron emission tomography | 6 months
  Regional myocardial perfusion below 2.3 ml/g/min measured by the quantitative positron emission tomography is a marker of myocardial ischemia
Presence of myocardial ischemia assessed by the cardiopulmanary exercise test | 6 months
  Criteria for myocardial ischemia that must be fulfilled are 1) Double sloping in the oxygen consumption/work rate trajectory, peak oxygen consumption below limit of the lowest normal, and abnormal oxygen pulse trajectory during the cardiopulmonary exercise test.

OTHER OUTCOMES:
Agreement in the detected myocardial ischemia between the myocardial perfusion positron emission tomography and the cardiopulmonary exercise testing | 6 months
  Positron emission tomography is the golden standard in the detection of myocardial ischemia. Results of cardiopulmary exercise testing will be compared with those of positron emission tomography using ROC-analysis. 6 months follow-up enables evaluation of reversibility of changes.

CONTACTS AND LOCATIONS:
Overall Officials: Tomi Laitinen, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio Univerity Hospital, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No